CLINICAL TRIAL: NCT00852670
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase IIa Study to Evaluate the Efficacy, Safety, and Tolerability of ACT-128800, an S1P1 Receptor Agonist, Administered for 6 Weeks to Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: ACT-128800 in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor, Actelion
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058A200
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — ponesimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: ACT-128800
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-128800 — ACT-128800 administered orally once daily
  Arms: A
Drug: Placebo — Matching placebo capsules administered orally once daily
  Arms: B

SUMMARY:
This study will assess the efficacy, safety, and tolerability of ACT-128800 in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females with moderate to severe plaque psoriasis who require systemic treatment and for whom participation in a placebo-controlled study of an investigational drug is justified.

Exclusion Criteria:

* Patients with other forms of psoriasis and patients who are currently treated for autoimmune disorders other than psoriasis.
* Systemic or topical treatments for psoriasis other than emollients.
* Ongoing bacterial, viral or fungal infections.
* History or presence of malignancy.
* Additional inclusion and exclusion criteria apply with respect to medical conditions and concomitant treatments which could affect patients' risk from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) percent change relative to baseline at Week 6 visit. | Baseline to week 6

SECONDARY OUTCOMES:
"Clear - almost clear" Physician Global Assessment (PGA) at Week 6 visit. | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Georg Schmidt, MD, Study Director — Actelion
Locations (14):
- Austria (2):
  - Landeskrankenhaus - Universitätsklilnikum Graz, Allgemeine Dermatologie, Graz
  - University Klinik of Vienna, Vienna
- France (3):
  - Departement de Pneumologie/ Unité Immunologie Clinique Allergie- Centre Hospitalier Lyon sud, Lyon
  - CHU de Nice-Hôpital de l'Archet 2 / Service de dermatologie, Nice
  - Dermatologie, Hôpital Purpan Universtité Paul Sabatier, Toulouse
- Germany (4):
  - Klinik für Dermatologie Venerologie und Allergologie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Department of Dermatology University Hospital Johannes Gutenberg-University Mainz, Mainz
  - University Clinic Münster Clinic and Policlinic for skin diseases, Münster
- Hungary (4):
  - Semmelweis Universtity Dept. dermato-venerology and skin oncology, Budapest
  - UNIVERSITY OF DEBRECEN Department of dermatology, Debrecen
  - University of Szeged Department of dermatology and allergology, Szeged
  - Veszprem County Csolnoky Ferenc Hospital Dermatology Department, Veszprém
- Clinical Centre of Nis Clinic of Dermato-venerology, Niš, Serbia